CLINICAL TRIAL: NCT02709642
Title: Brigham and Women's Healthy Weight Study: Randomized Controlled Trial of a Financial Incentive for Weight Maintenance
Brief Title: Brigham and Women's Healthy Weight Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1K23HL111211-03 (NIH)
Record Dates: First submitted 2016-03-08; First posted 2016-03-16 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Control Participants will complete weekly weigh-ins and receive emails about how their current weight compares to their baseline weight.
- Deposit Contract (Experimental): The deposit contract group will also complete weekly weigh-ins and receive emails about how their current weight compares to their baseline weight. In addition, the deposit contract group will be asked to make a deposit of at least $100 each 10-week period over the course of one year (50 weeks). Each week, they will recoup 1/10 of their 10-week deposit if they are within two pounds of their baseline weight or lower. If they are more than two pounds above their baseline weight, they will forfeit 1/10 of their 10-week deposit. The money they forfeited for that week will go into a collective pool to be divided up at the end of each 10-week period by all deposit contract participants who successfully maintained their weight loss at the end of the 10-week period.
  Interventions: Behavioral: Deposit Contract

INTERVENTIONS:
Behavioral: Deposit Contract — A deposit contract (DC) is an agreement in which study participants puts their own money at risk, with the goal of "earning" it back by achieving a goal, in this case maintaining prior weight loss. If DC participants successfully maintain their weight, they get their money back. If they are not successful, they lose their money. For each 10 week period for one year, DC participants will make a deposit of at least $100 but will be allowed to increase their contribution if they would prefer.
  Arms: Deposit Contract

SUMMARY:
The purpose of this study is to determine if a financial deposit contract is a successful method of helping people to maintain their weight loss. A deposit contract is an agreement in which participants put their own money at risk, with the goal of "earning" it back by achieving a goal, in this case maintaining prior weight loss. The study will also evaluate the interventions using survey research to assess the feasibility and acceptability of the interventions.

DETAILED DESCRIPTION:
Interested participants who can verify >10lb weight-loss over the last year and a half will be randomly assigned to either the control group, in which they will be asked to attend weekly weigh-ins at Brigham and Women's Hospital (BWH) over the course of a year, or to the deposit contract intervention group. Both the control group and the deposit contract group will complete the weekly weigh-ins for one year. The deposit contract group will additionally have a financial component: these participants will be asked to make a deposit of at least $100 each 10-week period over the course of one year (50 weeks), and can recoup this amount as detailed above. All participants will take baseline and end-of-study surveys.

During an enrollment meeting, study staff will request via an authorization form that participants allow approved members of the research staff to examine their electronic medical record for the duration of the study if they receive their care at a BWH-affiliated practice. This will confirm their >10lb weight loss.

At the end of every 10-week period, DC participants will receive an email with how much money they recouped. Participants who did not recoup the full amount they deposited must bring in a check to the following weigh-in to cover the difference so that participants have at least $100 deposited for the following 10-week period. Additionally, participants will have the option to use their initial study baseline weight, or be re-weighed for a new baseline weight for the following 10-week period, for which they will then use as their target weight. They will also have the option to increase or decrease their deposit for the upcoming 10-week period as needed.

Each subject may skip non-consecutive weigh-ins without losing their weekly contribution. However, if subjects skip two or more consecutive weekly weigh-ins, participants may only recoup up to one of those skipped weigh-ins if they are successful in their weight management in the week that they return for a weigh-in. Skipped weigh-ins will not roll over into a new 10-week period.

ELIGIBILITY:
Inclusion Criteria:

* employee of Brigham and Women's Hospital, Dana-Farber Cancer Institute (DFCI), Brigham and Women's Physicians Organization (BWPO), or Partners working at the Francis Street complex of Brigham and Women's Hospital (either part-time or full-time)
* 18 years of age or older
* successfully and intentionally lost at least 10lbs within the past 18 months
* had a BMI over 25 at some point over the previous 18 months

Exclusion Criteria:

* plan to change jobs outside of the BWH Francis Street complex in the next year
* had weight-loss surgery in the past 3 years
* currently on a very low calorie (800 or fewer calories) liquid diet or taking weight loss medicine
* currently have cancer, a severe psychiatric disorder, an eating disorder, or another severe medical illness that may affect weight beyond control
* plan to become pregnant in the next year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-06; Primary Completion 2018-07-01 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Weight | Weekly weigh-ins from baseline until the end of the study (about 1 year from April 2016-August 2017).
  Primary outcome measure will be the difference in weight in pounds between their baseline trial weight and their weight at 1 year, controlling for age, sex, race, and baseline weight.

SECONDARY OUTCOMES:
Success in meeting weight goal | Weekly weigh-ins from baseline until the end of the study (about 1 year from April 2016-August 2017).
  The binary variable of whether subjects met their goal at the end of one year will be assessed with logistic regression.
Number of weeks in which subjects met their weight goal | Weekly weigh-ins from baseline until the end of the study (about 1 year from April 2016-August 2017).
  The number of weeks in which subjects met their weight goal will be assessed with linear regression.
Number of participants who report factors of weight maintenance success as assessed by questionnaires | At Baseline (~April-August 2016) and at completion (~June-August 2017)
  Surveys at baseline and at follow-up will assess a variety of factors associated with weight maintenance, such as how participants have lost and are seeking to lose weight; how satisfied they are with their weight; their motivation and confidence in losing and maintaining weight loss; and behaviors such as diet, exercise habits, and screen time. These factors will be examined with basic descriptive statistics. Survey analysis will assess whether some of these factors, specifically confidence and motivation to lose or maintain weight, are associated with the primary outcome of weight change at 1 year, using linear regression models.

CONTACTS AND LOCATIONS:
Overall Officials: Jason P Block, MD, MPH, Principal Investigator — Obesity Prevention Program, Department of Population Medicine, Harvard Medical School, Harvard Pilgrim Health Care Institute, Boston, MA.
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available on a case-by-case basis.

REFERENCES:
- [Background] Volpp KG, John LK, Troxel AB, Norton L, Fassbender J, Loewenstein G. Financial incentive-based approaches for weight loss: a randomized trial. JAMA. 2008 Dec 10;300(22):2631-7. doi: 10.1001/jama.2008.804. PMID 19066383
- [Background] Jeffery RW, Thompson PD, Wing RR. Effects on weight reduction of strong monetary contracts for calorie restriction or weight loss. Behav Res Ther. 1978;16(5):363-9. doi: 10.1016/0005-7967(78)90005-0. No abstract available. PMID 743075